CLINICAL TRIAL: NCT05505708
Title: a Comparison Between the Effects of Crystalloids and Colloids on Lung Ultrasound Score in Preeclamptic Patients Undergoing Spinal Anesthesia for Caesarean Section: a Randomized Double Blinded Controlled Trial
Brief Title: a Comparison Between the Effects of Crystalloids and Colloids on Lung Ultrasound
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Karim mohamed abou elella, assisstant lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-76-2020
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema | interventions — Hydroxyethyl Starch Derivatives; Starch; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (V) (Active Comparator): Group (V): will receive hydroxyethyl starch (voluven) Pfizer Inc 500ml over 30 minutes
  Interventions: Drug: hydroxyethyl starch in sodium chloride injection Brand Name: Voluven
- Group (R) (Active Comparator): Group (R): will receive ringer acetate 500ml over 30 minutes
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: hydroxyethyl starch in sodium chloride injection Brand Name: Voluven — (6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride injection) is a clear to slightly opalescent, colorless to slightly yellow, sterile, non-pyrogenic, isotonic solution for intravenous administration using sterile equipment.
  Each 100 mL of the solution contains: 6 g of Hydroxyethyl Starch 130/0.4 and 900 mg of Sodium Chloride USP in Water for Injection USP.
  In addition, sodium hydroxide, USP, or Hydrochloric acid, USP, has been added to adjust the final pH so the final solution pH is 4.0 to 5.5.
  Other Names: starch
  Arms: Group (V)
Drug: saline solution — Within each 100 mL of 0.9% sodium chloride Injection USP, there is 15.4 mEq of sodium ions and 15.4 mEq of chloride ions. Additionally, the osmolarity is 308 mOsmol/liter, and it has a pH range of 4.5 to 7
  Other Names: normal saline
  Arms: Group (R)

SUMMARY:
This study is designed to compare the effect of crystalloids and colloids on lung ultrasound score in preeclapmtic pregnant cases undergoing spinal anesthesia for caesarean section

Objectives:

To identify ideal fluid in order to maintain proper intravascular volume in preeclamptic patients that allows organ perfusion without causing lung congestion or pulmonary edema

Hypothesis:

the investigators hypothesize that colloids are better than crystalloids in maintaining good intravascular volume without affecting lung ultrasound score.

DETAILED DESCRIPTION:
Hypertensive disorders are the most common complications of pregnancy. They occur in 6-8% of pregnancies and account for approximately 15% of maternal deaths in the United States Pre-eclampsia is a pregnancy-specific syndrome of unknown etiology that is defined as systolic blood pressure (SBP) > 140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg presenting after 20 weeks of gestation with significant proteinuria (1) Because patients with pre-eclampsia may have significant intravascular volume deficit and reduced uteroplacental perfusion, it is prudent to administer fluids before any anesthetic interventions. (2) however it may increase their risk of developing pulmonary oedema (3) Colloids and crystalloids are two types of fluids that are used for fluid replacement, as volume expanders. Crystalloids are low-cost salt solutions (e.g. saline) with small molecules, which can move around easily when injected into the body. Colloids can be man-made (e.g. starches, dextrans, or gelatins), or naturally occurring (e.g. albumin or fresh frozen plasma (FFP)), and have bigger molecules, so stay in the blood for longer before passing to other parts of the body. (4) Women with pre-eclampsia lose protein through renal excretion and may also extravasate protein into the interstitial tissues, oncotic pressure falls because of this and the tendency to lose fluid from the intravascular space is partially determined by this mechanism. Filling the vascular space with fluid will lead to increasing peripheral oedema. Colloids will remain in the vascular compartment for longer periods than crystalloids although the loss of colloid into the interstitial tissues will also contribute to the development of oedema. Changes in capillary permeability will have an independent influence. (5) Ultrasound is now widely used in many medical specialties, being safe tool for both the parturient and the baby, ultrasound is basically used by the obstetricians in pregnant females for diagnosis of fetal presentation, placental position, fetal organs, amount of liquor and in some interventions amniocentesis. In the last 15 years, a new imaging application of sonography has emerged in the clinical arena: lung ultrasound (LUS), it can give valuable data in diagnosing and management of pneumothorax, pleural effusion, lung consolidation and pulmonary congestion. (6) The electrical cardiometry which can be used to measure and calculate hemodynamic parameters such as cardiac output, stroke volume, systemic vascular resistance, ICON (index of contractility), and thoracic fluid content. (7) In general, there is no epidemiological evidence to support the choice of colloidal solutions over crystalloids and it is not clear that colloidal solutions would be more effective and less likely to cause harm than crystalloids in preeclamptic patients. A meta-analysis was done to investigate crystalloid versus colloid resuscitation in critically ill patients however pregnant women and neonates were excluded. (8) Consequently, there is inadequate evidence supporting one view or another in the management of pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant cases with preeclampsia: gestational age >32 weeks
2. Singleton pregnancy
3. Age above 18 years

Exclusion Criteria:

1. Pregnant cases with preeclampsia: gestational age >32 weeks
2. Singleton pregnancy
3. Age above 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2022-12-05 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
changes in Lung ultrasound score | changes in lung ulrasound is measured by comparing the alvelo interstitial score at baseline (before ) receiving spinal anaesthesia then after 30 minutes
  Alveolo-interstitial syndrome is assessed by the measurement of multiple B-lines

CONTACTS AND LOCATIONS:
Overall Officials: abd elbar, MD, Principal Investigator — kasr alainy hospital
Locations (1):
- Kasr Elainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested
Supporting Information: Study Protocol, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact clinicalresearchsupportcenter@ucdenver.edu."
URL: http://clinicalresearchsupportcenter@ucdenver.edu